CLINICAL TRIAL: NCT04132479
Title: Sequential Helicobacter Pylori Eradication Therapy in Myanmar; a Randomized Clinical Trial of Efficacy and Tolerability
Brief Title: The Epidemiology and Optimal Treatment of Helicobacter Pylori in Myanmar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: University of Medicine 2, Yangon, Myanmar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC17980
Record Dates: First submitted 2019-09-15; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Clarithromycin; Amoxicillin; Tinidazole; Rabeprazole

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequential therapy (Experimental): Sequential Clarithromycin + Amoxycillin + Tinidazole + rabeprazole by mouth (Both amoxycillin 1000mg every 12 hours and rabeprazole 20 mg every 12 hours for 5 days, followed by clarithromycin 500 mg every 12 hours, tinidazole 500mg every 12 hours and rabeprazole 20 mg every 12 hours for 5 days)
  Interventions: Drug: Clarithromycin 500mg; Drug: Amoxicillin 500mg; Drug: Tinidazole 500mg; Drug: Rabeprazole 20mg
- Concomitant therapy (Active Comparator): Concomitant clarithromycin 500mg every 12 hours + amoxycillin 1000mg every 12 hours + tinidazole 500mg every 12 hours + rabeprazole 20mg every 12 hours (all drugs by mouth for 14 days).
  Interventions: Drug: Clarithromycin 500mg; Drug: Amoxicillin 500mg; Drug: Tinidazole 500mg; Drug: Rabeprazole 20mg

INTERVENTIONS:
Drug: Clarithromycin 500mg — 1000mg taken orally every 12 hours for 5 days
  Other Names: Getz Pharma, Karachi, Pakistan
  Arms: Sequential therapy
Drug: Amoxicillin 500mg — 1000mg taken orally every 12 hours for 5 days
  Other Names: Denk Pharma, Munich, Germany
  Arms: Sequential therapy
Drug: Tinidazole 500mg — 500mg taken orally every 12 hours for 5 days
  Other Names: Global Pharma, Chennai, India
  Arms: Sequential therapy
Drug: Rabeprazole 20mg — 20mg taken orally every 12 hours for 5 days
  Other Names: Zifam Pinnacle, Mumbai, India
  Arms: Sequential therapy
Drug: Clarithromycin 500mg — 1000mg taken orally every 12 hours for 14 days
  Other Names: Getz Pharma, Karachi, Pakistan
  Arms: Concomitant therapy
Drug: Amoxicillin 500mg — 1000mg taken orally every 12 hours for 14 days
  Other Names: Denk Pharma, Munich, Germany
  Arms: Concomitant therapy
Drug: Tinidazole 500mg — 500mg taken orally every 12 hours for 14 days
  Other Names: Global Pharma, Chennai, India
  Arms: Concomitant therapy
Drug: Rabeprazole 20mg — 20mg taken orally every 12 hours for 14 days
  Other Names: Zifam Pinnacle, Mumbai, India
  Arms: Concomitant therapy

SUMMARY:
This study aims to:

1. Determine the prevalence of Helicobacter infection in Myanmar (this would be the largest ever series in the country)
2. Determine the clinical and epidemiological associations of Helicobacter infection in Myanmar
3. Determine the utility of stool antigen testing to diagnose the infection and confirm eradication
4. Compare the relative efficacies of concomitant and sequential therapy
5. Determine the relative efficacies of first, second and third line therapies in Myanmar in 2018

DETAILED DESCRIPTION:
There are very few published studies to examine the prevalence of Helicobacter infection in Myanmar. Two previous studies (both < 400 participants) suggested that the prevalence was approximately 50% (Myint WJG 2015, Aye MMJ 2015).

The high prevalence of H.pylori is important because gastric adenocarcinoma is the fourth most common cancer in the country (WHO 2014). Gastric cancer has an almost uniformly dismal 5-year survival rates in this resource-limited country and is estimated to kill almost 5000 patients per year in Myanmar (WHO 2014).

In addition, anecdotally there is a significant associated burden of peptic ulcer disease in the country, although there are few published data to examine the issue.

Strategies to diagnose and eradicate H.pylori must be considered in the context that the annual per capita health budget is USD103 (World Bank 2016).

Therapeutic regimens must also consider the issue of antimicrobial resistance, which varies from country to country. There are very few data from Myanmar to guide us and those that are available vary enormously.

In vitro antibiotic resistance by agent

Amoxycillin 0%, 8%, 7%

Metronidazole 33%, 54%,100%

Clarithromycin 0%, 13%, 50%

Levofloxacin 6%, NR, 3%

Tetracycline 0%, NR, NR

Ciprofloxacin 6%, NR NR

Studies: Mahachai 2012, Aye 2005, Aye 2014

However, it is also known that in vitro resistance does not necessarily translate into in vivo failure. Furthermore in a resource poor setting like Myanmar, a strategy of susceptibility guided treatment is not feasible. Indeed, this is not likely to be cost-effective in even wealthy countries (ACG guidelines 2017 and Maastricht consensus guidelines 2017).

The current first line therapy for H.pylori in Myanmar is 10-14 days of concomitant bd PPI + bd Clarithromycin + bd Amoxycillin + bd metronidazole. This regimen contains up to 126 pills (14 days) and costs up to USD16 (14 days). It is likely that 14 days of 4 drug therapy will generate issues with side effects and adherence, although again this has not been examined locally.

Alternatively, a 10-day sequential regimen of 5 days of bd PPI + Amoxycillin, then 5 days of bd PPI + Clarithromycin and Tinidazole reduces the pill load to 50 pills and the total drug cost to USD6. This regimen has been shown to be highly effective in Slovenia (94.2%), Portugal (90%), Belgium (90%), Israel (95.9%), Thailand (94%), Taiwan (91.9%), Singapore (90.3%), and the United Arab Emirates (88.6%) (Review, De Francesco 2017).

A sequential regimen has been shown to have less satisfactory success rates in Greece , Spain, Ireland, Turkey, Iran, Korea, China, and Puerto Rico (although in many of these studies, metronidazole was used instead of tinidazole (Review, De Francesco 2017)).

The current second-line regimen in Myanmar is 10-14 days of bd PPI + Levofloxacin + Amoxycillin (pill load 80 pills for 10 days, total cost USD3). In this era of evolving drug resistance, we may not want to use quinolones as first line therapy however.

The current third line therapy is Bismuth based quadruple therapy (BQT). This regimen is comprised of Bismuth + PPI + Tetracycline + Tinidazole (pill load 120 pills, total cost USD50)

The proposed study aims to demonstrate that a 10-day course of sequential therapy is not inferior to 14 days of 4 drug concomitant therapy. Assuming a cure rate of 80% for Concomitant 4 drug therapy, and an inferiority bound of 10%, the sample size is 626 (313 patients in each arm). To identify 626 patients, we will need to screen approximately 1250 patients. In this resource-poor setting, diagnosis will be established using monoclonal stool antigen testing (SAT BioMerieux BioNexia). Patients who test positive with SAT will be randomised 1:1 in an open label study to either a 10-day course of sequential therapy or the current first line regimen of concomitant 4 drug therapy. Four weeks after completing therapy, eradication will be confirmed with repeat SAT.

Those patients failing the first line therapy would then receive second line levofloxacin and then tested to confirm eradication. This would determine the efficacy of the country's current second line therapy.

Finally, patients failing first and second line therapy would receive the more involved and expensive third line therapy. Once again, this would determine the efficacy of third line therapy.

To ensure all participants had their H.pylori infection eradicated, those failing three lines of therapy would be offered endoscopy and culture directed therapy.

The performance of the stool antigen test is affected by the PPI therapy, so the study can't easily enrol patients presenting with acute symptoms who will frequently have already been taking PPI therapy (higher rate of false negatives). Therefore, the study will enrol outpatients about to commence aspirin, NSAIDs or anticoagulants (in whom the risk of GI bleeding is higher) or patients with a personal history of peptic ulcer disease or family history of gastric cancer. These are all indications for H.pylori testing (ACG guidelines 2017 and Maastricht consensus guidelines 2017).

Outputs

1. The prevalence of H.pylori in Yangon, Myanmar
2. Clinical and demographic associations of H.pylori infection in Myanmar
3. Efficacy of

   1. Current first line therapy: 14 days of concomitant PPI + amoxy + clari + metro
   2. Alternative: 10 days of sequential PPI + amoxy + clari + Tinidazole
   3. Current second line therapy: 14 days of PPI + Levo + Amoxy
   4. Current third line therapy: 14 days of Bismuth + PPI + tetracycline + metro (BQT)
4. Acceptability - to patients and staff - of stool antigen testing for H.pylori screening and for confirming eradication.

ELIGIBILITY:
Inclusion Criteria:

* Satisfies one of the criteria for H. pylori testing in the 2017 American College of Gastroenterology guidelines
* Informed consent

Exclusion Criteria:

* No informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of sequential Helicobacter Pylori Eradication Therapy versus concomitant Helicobacter Pylori Eradication Therapy. | 4 weeks after completion of initial eradication therapy, at an average of 6 weeks after randomization.
  The proportion of participants with a negative stool antigen test 4 weeks after end of treatment in those who received Sequential Helicobacter Pylori Eradication Therapy compared with those who received concomitant Helicobacter Pylori Eradication Therapy.

SECONDARY OUTCOMES:
The number of participants with adverse drug reactions | During therapy with the agents and follow up for the 4 weeks after completion of antibiotic therapy; a total of 6 weeks.
  Participants will be reviewed as outpatients in face-to-face interviews on days 5, 11 and 15 where the number of participants with treatment-related adverse events will be recorded. Patients will also be reviewed when they return for testing to confirm eradication.
  The study pro forma will prompt clinicians to ask specifically about the presence or absence of the following gastrointestinal side effects: vomiting, nausea, diarrhoea and abdominal discomfort and the following systemic side effects: dizziness and headache. If the participants have any other symptoms that they feel are related to the medication, these will also be recorded.
  The presence or absence of each individual side effect and the total number of side effects experienced by participants in the two arms will be compared. The severity of each side effect will not be quantified.
Adherence to therapy | 14 days
  Participants will be reviewed as outpatients in face-to-face interviews on days 5, 11 and 15 where a pill count will be performed to assess adherence using the 4 item Morisky Medication Adherence Scale (MMAS-4, minimum value 0, maximum value 4, the higher score the better the adherence)

OTHER OUTCOMES:
Loss to follow up | Through study completion, an average of 3 months
  The number of participants lost to follow up defined as a failure to attend follow appointment and an inability to be contacted by telephone on 3 separate occasions.
Mortality | Through study completion, an average of 3 months
  The rate and cause of death among participants

CONTACTS AND LOCATIONS:
Overall Officials: Mar Mar Kyi, MD, Study Chair — University of Medicine 2, Yangon, Myanmar
Locations (1):
- Insein General Hospital, Yangon, Burma

IPD SHARING:
Plan to Share IPD: No